CLINICAL TRIAL: NCT02017145
Title: Role of Post-operative Re-application of Chloraprep® Following Lower Extremity Surgeries on Surgical Site Bacterial Colonization.
Brief Title: Study on the Reapplication of Chloraprep After Lower Extremity Surgery and Prior to Dressing Application
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sanford Health (Other)
Responsible Party: Principal Investigator, Kyle Judd, Employed Physician, Sanford Health
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SH Chloraprep reapplication
Record Dates: First submitted 2013-12-16; First posted 2013-12-20 (Estimated); Last update posted 2014-02-19 (Estimated); Status verified 2014-02

CONDITIONS: Lower Extremity Surgery; Surgical Site Infection; Bacterial Colonization; Surgical Antiseptic
Keywords: infection; chloraprep; chlorhexidine; lower extremity surgery; antiseptic; bacterial colonization
MeSH Terms: conditions — Surgical Wound Infection; Infections

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- no reapplication (No Intervention): This group will not have chloraprep reapplied after their surgery and prior to dressing application.
- reapplication (Experimental): This group will have chloraprep reapplied following their lower extremity surgical procedure and prior to dressing application.
  Interventions: Drug: Chloraprep

INTERVENTIONS:
Drug: Chloraprep
  Arms: reapplication

SUMMARY:
The purpose of the current work is to determine the efficacy of the re-application of surgical prep solution in decreasing surgical site bacterial contamination following lower extremity surgery. Decreasing the extent of bacterial colonization of the skin surrounding the surgical site during the initial healing phases would theoretically decrease the rate of infection in high-risk persons.

ELIGIBILITY:
Inclusion Criteria:

* Male and female
* Adults (18+)
* Both elective and non-elective procedures
* Lower extremity surgery performed below the knee and requiring post-operative splint immobilization for 2-3 weeks
* Able to understand and read the English language
* Signed informed consent

Exclusion Criteria:

* Pregnant (to be assessed the day of surgery per standard of care surgical protocol)
* Known allergies to chlorhexidine gluconate or isopropyl alcohol
* Multiple planned lower extremity surgeries
* Local skin disease
* Pre-existing or known infection at surgical site
* Open wounds or local abrasions
* Unable to or unwilling to follow through with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2014-02; Primary Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
quantitative bacterial colonization | 14-21 days
  Compare the number of colony forming units taken from culture swabs immediately adjacent to the wound during dressing change between the two arms
positive culture rate | 14-21 days
  Compare the overall positive culture rate between the two treatment groups

SECONDARY OUTCOMES:
bacterial strain identification | 14-21 days
  Assess the total number of bacterial strains and identifying those strains cultured from swabs taken immediately adjacent to the wound during dressing change

CONTACTS AND LOCATIONS:
Overall Officials: Kyle T Judd, MD, Principal Investigator — Sanford Orthopedics and Sports Medicine
Locations (1):
- Sanford USD Medical Center, Sioux Falls, South Dakota, United States

REFERENCES:
- [Background] Gould D. Causes, prevention and management of surgical site infection. Nurs Stand. 2012 Jul 25-31;26(47):47-56; quiz 58. doi: 10.7748/ns2012.07.26.47.47.c9226. PMID 22913092
- [Background] Ostrander RV, Botte MJ, Brage ME. Efficacy of surgical preparation solutions in foot and ankle surgery. J Bone Joint Surg Am. 2005 May;87(5):980-5. doi: 10.2106/JBJS.D.01977. PMID 15866959
- [Background] Darouiche RO, Wall MJ Jr, Itani KM, Otterson MF, Webb AL, Carrick MM, Miller HJ, Awad SS, Crosby CT, Mosier MC, Alsharif A, Berger DH. Chlorhexidine-Alcohol versus Povidone-Iodine for Surgical-Site Antisepsis. N Engl J Med. 2010 Jan 7;362(1):18-26. doi: 10.1056/NEJMoa0810988. PMID 20054046
- [Background] Hibbard JS. Analyses comparing the antimicrobial activity and safety of current antiseptic agents: a review. J Infus Nurs. 2005 May-Jun;28(3):194-207. doi: 10.1097/00129804-200505000-00008. PMID 15912075
- [Background] Hibbard JS, Mulberry GK, Brady AR. A clinical study comparing the skin antisepsis and safety of ChloraPrep, 70% isopropyl alcohol, and 2% aqueous chlorhexidine. J Infus Nurs. 2002 Jul-Aug;25(4):244-9. doi: 10.1097/00129804-200207000-00007. PMID 12131506